CLINICAL TRIAL: NCT03358680
Title: Temperature and Analgesia Monitoring During Cardial Parmonary Bypass
Status: Completed | Type: Observational
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Other Study IDs: ZYLX201706-11025
Record Dates: First submitted 2017-11-13; First posted 2017-11-30 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: noninvasive analgesia measurement — noninvasive analgesia measurement using index of consciousness(IOC2)
  Other Names: index of consciousness(IOC2)

SUMMARY:
1. Investigator will apply IOC2 to reflect the depth of analgesic during hypothermia in CPB period.
2. effectiveness of IOC2 monitoring for anesthetic depth versus commonly used vital sign monitoring based on factors such as blood pressure and heart rate.
3. Evaluate the other sedation co-relation measurement, include BIS , IOC2 to reflected the consciousness during the operation.
4. Evaluate the other hemodynamic index, include CO, SVV, CVP, PPV to reflect the circulation function , and the effect to the IOC2 and IOC1.
5. Describe the trend of all the measurement. detect the variation of the index during the temperature change during the CPB.

DETAILED DESCRIPTION:
In this study,

1. Investigator will apply IOC2 to reflect the depth of analgesic during hypothermia in CPB period.
2. Furthermore, investigator evaluated the effectiveness of IOC2 monitoring for anesthetic depth versus commonly used vital sign monitoring based on factors such as blood pressure and heart rate.
3. Evaluate the other sedation co-relation measurement, include BIS , IOC2 to reflected the consciousness during the operation.
4. Evaluate the other hemodynamic index, include CO, SVV, CVP, PPV to reflect the circulation function , and the effect to the IOC2 and IOC1.
5. Describe the trend of all the measurement. detect the variation of the index during the temperature change during the CPB.

ELIGIBILITY:
Inclusion Criteria:

* undergoing coronary artery bypass surgery

Exclusion Criteria:

* change the surgery planning during the operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients schedule undergoing coronary artery bypass surgery
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
IOC2 | 1 DAY
  Index of consciousness 2

SECONDARY OUTCOMES:
BIS | 1 DAY
  to monitor and compare appropriate conscious value
IOC1 | 1 DAY
  index of consciousness 1

CONTACTS AND LOCATIONS:
Overall Officials: Zhaolong Tian, MS, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China